CLINICAL TRIAL: NCT02640612
Title: Long-term Assessment of Safety, Efficacy, Pharmacokinetics and Immunogenicity of BI 695501 in Patients With Rheumatoid Arthritis (RA): an Open-label Extension Trial for Patients Who Have Completed Trial 1297.2 and Are Eligible for Long-term Treatment With Adalimumab
Brief Title: Long-term Assessment of Safety and Efficacy of BI 695501 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1297.3; 2015-002634-41 (EudraCT Number)
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — BI 695501

ARMS (1):
- BI 695501 (Experimental)
  Interventions: Drug: BI 695501

INTERVENTIONS:
Drug: BI 695501

SUMMARY:
The main objective of this trial is to provide long-term safety, pharmacokinetics (PK), and immunogenicity data on BI 695501 administered via prefilled syringe in patients with Rheumatoid Arthritis who have completed Trial 1297.2. The primary endpoint thereby is the number (proportion) of patients with drug-related adverse events (AEs) during the treatment phase. The secondary objective in this trial is the assessment of Long-term efficacy of BI 695501 by evaluation of:

* the change from Baseline in DAS28 (ESR) at Week 48
* the proportion of patients meeting American College of Rheumatology 20% (ACR20) response criteria at Week 48
* the proportion of patients who meet the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) definition of remission at Week 48
* the proportion of patients with EULAR response (good response, moderate response, or no response) at Week 48.

ELIGIBILITY:
Inclusion criteria:

* All patients must sign and date an Informed Consent Form consistent withInternational Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines and local legislation prior to participation in the trial (i.e., prior to any trial procedures, which include medication washout and restrictions) and be willing to follow the protocol.
* Adult patients with moderately to severely active RA who have completed Trial 1297.2, and who wish to participate in this extension trial and in the investigator´s assessment can benefit from receiving BI 695501.
* Patients willing and able to self-administer BI 695501 pre-filled syringe.
* Willing to use a reliable means of contraception throughout trial participation (females) and willing to use an acceptable method of contraception for 6 months following completion or discontinuation from the trial medication males and females).

Exclusion criteria:

* Investigator-reported drug-related Serious Adverse Events (SAEs) in Trial 1297.2
* ACR functional Class IV or wheelchair/bed bound
* Primary or secondary immunodeficiency (history of, or currently active)
* Positive QuantiFERON test
* Known clinically significant coronary artery disease or significant cardiac arrhythmias or severe congestive heart failure (NYHA Classes III / IV), or interstitial lung disease
* Anaphylactic reaction or hypersensitivity to adalimumab in Trial 1297.2
* History / recent evidence of cancer incl. solid tumours, hematologic malignancies, and carcinoma in situ (certain exceptions permitted)
* Positive serology for Hepatitis B virus (HBV) or Hepatitis C virus (HCV)
* Planned live virus or bacterial vaccinations during the trial, or up to 3 months after the last dose of trial drug
* Receipt or treatment (including biologic therapies) that may place the patient at unacceptable risk during the trial
* Significant disease (disease which may (i) put the patient at risk because of participation or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial) other than RA and/or a significant uncontrolled disease
* Women: premenopausal (last menstruation 1 year prior to screening), sexually active, pregnant or nursing, or of child-bearing potential and not practicing an acceptable method of birth control, or not planning to use an acceptable method of birth control throughout the trial
* Current inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, etc.) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, pulmonary fibrosis, etc.). Secondary Sjögren´s syndrome or secondary limited cutaneous vasculitis with RA is permitted
* Any planned surgical procedure, including bone/joint surgery/synovectomy for the duration of the trial
* Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with iv. anti-infectives within 4 weeks of the Screening Visit or completion of oral anti-infectives within 2 weeks of the Screening Visit
* Serious infection or opportunistic infection during the 1297.2 trial
* Any acquired neurological, vascular, systemic or demyelinating disorder that might affect any of the efficacy assessments, in particular, joint pain and swelling (e.g., Parkinson´s disease, cerebral palsy, diabetic neuropathy) that occurred during the 1297.2 trial.
* Currently active alcohol or drug abuse
* Treatment with iv. Gamma Globulin or the Prosorba® Column during the 1297.2 trial
* Planned treatment with iv. intramuscular, intra-articular and parenteral corticosteroids
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >1.5 times upper limit of normal (ULN)
* Hemoglobin <8.0 g/dL
* Platelets <100,000/µL
* Leukocyte count <4000/µL
* Creatine clearance <60 mL/min
* Current participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (89):
- United States (29):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - TriWest Research Associates, LLC, El Cajon, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Science and Research Institute, Inc., Jupiter, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Lovelace Scientific Resources, Incorporated, Venice, Florida
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Arthritis Education and Treatment Center, Grand Rapids, Michigan
  - Accurate Clinical Research, Inc., Lincoln, Nebraska
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - STAT Research, Incorporated, Dayton, Ohio
  - Clinical Research Source, Inc., Toledo, Ohio
  - Center for Inflammatory Disease, Nashville, Tennessee
  - Adriana Pop Moody Clinic PA, Corpus Christi, Texas
  - Accurate Clinical Management LLC, Houston, Texas
  - Accurate Clinical Research, Incorporated, Houston, Texas
  - Rheumatology Clinic Of Houston, P.A., Houston, Texas
  - Arthritis & Osteoporosis Associates LLP, Lubbock, Texas
  - Heartland Research Associates, LLC, San Antonio, Texas
  - Danville Orthopedic Clinic, Incorporated, Danville, Virginia
  - Arthritis Northwest, PLLC, Spokane, Washington
- Bulgaria (9):
  - MHAT "Eurohospital" - Plovdiv, OOD, Plovdiv
  - MHAT "Trimontium", OOD, Plovdiv, Plovdiv
  - MHAT - Kaspela, EOOD, Plovdiv
  - Medical Center "Teodora", EOOD, Ruse, Rousse
  - MHAT,Fourth Dept. of Therapeutics & Cardiology, Ruse, Rousse
  - MHAT Shumen AD, Shumen, Shumen
  - MMA HAT Sofia, Bulgaria, Sofia
  - UMHAT Sv. Ivan Rilski EAD, Sofia
  - MDHAT 'Dr. Stefan Cherkezov', AD, Veliko Tarnovo
- Chile (5):
  - Corporacion de Beneficencia Osorno, Osorno
  - Quantum Research Santiago, Puerto Varas, Puerto Varas
  - Centro Medico Prosalud, Santiago
  - BIOMEDICA, Santiago, Santiago
  - CINVEC - Centro de Investigacion Clinica V Reg.,Vina del Mar, Viña del Mar
- Estonia (2):
  - Pärnu Hospital, Pärnu, Pärnu
  - Medita Kliinik OÜ, Tartu, Tartu
- Rheumazentrum Prof. Dr. G. Neeck, Bad Doberan, Bad Doberan, Germany
- Hungary (2):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klin. Kozpont, Szeged
  - Csolnoky Ferenc Korhaz, Veszprem, Veszprém
- Malaysia (2):
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Pulau Pinang, Pulau Pinang
- Poland (12):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Medica Pro Familia Spolka Akcyjna, Oddzial w Gdyni, Gdynia
  - MCBK Iwona Czajkowska Anna Podrazka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Medical Centre Pratia Katowice I, Katowice
  - Medical Centre Pratia Krakow, Krakow
  - Specialist Center ALL-MED, Krakow, Krakow
  - Niepubliczny ZOZ, "Nasz Lekarz", Lekarzy Rodzinnych z, Torun
  - Medical Centre Pratia Warszawa, Warsaw
  - Reumatika, Rheumatology Center, non-public outpatient clinic, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
- Russia (7):
  - Kemerovo SMA b/o War Veterans Regional Clinical Hospital, Kemerovo
  - Practicheskaya Meditsina Ltd, Moscow
  - Republic Kareliya Republican Hosp. named after V.A. Baranov, Petrozavodsk
  - Samara Regional Clinical Hospital n.a MI Kalinin, Samara, Samara
  - Stavropol State Medical Academy, Stavropol
  - Emergency Clinical Hospital n. a. N. V. Solovyev, Yaroslavl, Yaroslavl
  - SBHI of Yaroslavl Area "Clinical Hospital #3", Yaroslavl
- Serbia (4):
  - Institute of Rheumatology, Belgrade, Belgrade
  - Institute for Treatment and Rehabilitation, Niska Banja, Niška Banja
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital "Dr Laza K. Lazarevic" Sabac, Sabac, Šabac
- South Korea (2):
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital Universitario de Cruces, Barakaldo
  - Hosp. Nuestra Señora de la Esperanza, Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico de Santiago, Santiago de Compostela
- Siriraj Hospital, Bangkok, Thailand
- Ukraine (10):
  - Ivano-Frankivsk Nat. Medical University, Dept. Endocrinology, Ivano-Frankivsk
  - L.T. Malaya Institute of Therapy AMS of Ukraine, Kharkiv
  - CI of Healthcare Kharkiv CCH #8, Kharkiv, Kharkiv
  - SI NSC M.D. Strazhesko Institute Cardiology of NAMSU, Kyiv, Kyiv
  - Kjiv City Oleksandrivska Clinical Hospital, Kyiv
  - SI D.F.Chebotariov Institute of Gerontology of NAMSU, Kyiv, Kyiv
  - M.V. Sklifosovskyi Poltava RCH, Poltava, Poltava
  - M.I. Pyrogov VRCH, Vinnytsia, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia, Vinnytsia
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia, Zaporizhzhia

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Kang J, Eudy-Byrne RJ, Mondick J, Knebel W, Jayadeva G, Liesenfeld KH. Population pharmacokinetics of adalimumab biosimilar adalimumab-adbm and reference product in healthy subjects and patients with rheumatoid arthritis to assess pharmacokinetic similarity. Br J Clin Pharmacol. 2020 Nov;86(11):2274-2285. doi: 10.1111/bcp.14330. Epub 2020 Jun 11. PMID 32363771
- [Derived] Cohen SB, Czeloth N, Lee E, Klimiuk PA, Peter N, Jayadeva G. Long-term safety, efficacy, and immunogenicity of adalimumab biosimilar BI 695501 and adalimumab reference product in patients with moderately-to-severely active rheumatoid arthritis: results from a phase 3b extension study (VOLTAIRE-RAext). Expert Opin Biol Ther. 2019 Oct;19(10):1097-1105. doi: 10.1080/14712598.2019.1645114. Epub 2019 Aug 6. PMID 31387417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an open-label extension trial. Adult patients with moderate to severely active rheumatoid arthritis (RA) who completed Trial NCT02137226 (1297.2), wished to participate in this extension trial and per Investigator's assessment could benefit from continuing to receive BI 695501 were included in this trial.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. The screening visit of this trial was the Week 48 visit in Trial 1297.2.
Groups:
- BI 695501 to BI 695501: Patients initially randomized to BI 695501 in Period 1 and re-randomized to BI 695501 in Period 2 of the 1297.2 trial. Each patient received 40 milligram (mg)/0.8 millilitre (mL) BI 695501 in period 1 and 40 mg/0.8 mL BI 695501 in period 2. The respective treatment was administered by subcutaneous (SC) injection every 2 weeks from Day 1 to Week 48.
- Humira® to Humira®: Patients initially randomized to Humira® in Period 1 and re-randomized to Humira® in Period 2 of the 1297.2 trial. Each patient received 40 mg/0.8 mL Humira® in period 1 and 40 mg/0.8 mL Humira® in period 2. The respective treatment was administered by SC injection every 2 weeks from Day 1 to Week 48.
- Humira® to BI 695501: Patients initially randomized to Humira® in Period 1 and re- randomized to BI 695501 in Period 2 of the 1297.2 trial. Each patient received 40 mg/0.8 mL Humira® in period 1 and 40 mg/0.8 mL BI 695501 in period 2. The respective treatment was administered by SC injection every 2 weeks from Day 1 to Week 48.
Period: Overall Study
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
Started | 225 | 103 | 102
Completed | 203 | 89 | 96
Not Completed | 22 | 14 | 6
Not completed — Adverse Event | 6 | 7 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 3 | 3
Not completed — Lost to Follow-up | 4 | 1 | 1
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): All patients who received at least 1 dose during trial 1297.3. In the event of doubt as to whether a patient was treated or not, they were assumed to have been treated for the purposes of analysis, and thus included in the SAF. Patients were classified according to randomized/re-randomized treatments of Trial 1297.2.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501 | Total
Number analyzed (Participants) | 225 | 103 | 102 | 430
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of all patients included in the trial Population: SAF
  Years | 53.8 (11.87) | 51.7 (11.21) | 54.6 (9.90) | 53.5 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution of all patients included in the trial. Population: SAF
  Participants
    Female | 188 | 88 | 84 | 360
    Male | 37 | 15 | 18 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of all patients included in the trial Population: SAF
  Participants
    Hispanic or Latino | 23 | 8 | 10 | 41
    Not Hispanic or Latino | 199 | 94 | 92 | 385
    Unknown or Not Reported | 3 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of all patients included in the trial Population: SAF
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 7 | 2 | 0 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 0 | 2 | 5
    White | 215 | 100 | 100 | 415
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Drug-related Adverse Events (AEs) During the Treatment Phase
Description: The analysis of AEs was based on the concept of treatment-emergent AEs (TEAEs). Thus, all AEs with an onset after the first dose of trial drug up to a period of ten weeks after the last dose of trial drug were assigned to the current treatment for evaluation. Investigator assessed drug related AEs were AEs with a relationship to drug ticked "yes" according to the Investigator.
Time Frame: From the first drug administration until 10 weeks after the last drug administration, up to 58 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
Number analyzed (Participants) | 225 | 103 | 102
Percentage of patients (%) | 21.3 | 20.4 | 17.6

2. Secondary Outcome: Change From Baseline in Disease Activity Score in 28 Joints (DAS 28) by Erythrocyte Sedimentation Rate (ESR) at Week 48
Description: The DAS28 (ESR) score was derived using the following formulae: DAS28 (ESR) = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.014*(GH) + 0.7*ln(ESR) Where: • TJC28 = 28 joint count for tenderness • SJC28 = 28 joint count for swelling • GH = General Health component of the DAS (patient's global assessment of disease activity) • Ln (ESR) = natural logarithm of ESR. Last observation carried forward (LOCF) is the method used for handling missing components post baseline. Baseline for this trial was taken from the baseline of 1297.2. Improvement in DAS28 was also categorized using the European League Against Rheumatism (EULAR) response criteria. The DAS28 provides a number on a scale from 0 to 10 where higher values mean a higher disease activity. A DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
Time Frame: Baseline and Week 48.
Population: FullAnalysisSet(FAS) includes patients from the all subjects assigned set who received at least 1 dose of trial drug in Trial 1297.3 and had at least 1 DAS28(ESR and C-reactive protein) or american college of rheumatology 20% response criteria (ACR20) measured during trial. Classified according to randomized/rerandomized treatments of trial 1297.2.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
Number analyzed (Participants) | 225 | 103 | 101
Unit on scale | -3.01 (1.385) | -2.91 (1.323) | -2.98 (1.218)

3. Secondary Outcome: Percentage of Patients Meeting American College of Rheumatology (ACR) 20% Response Criteria at Week 48
Description: The proportion of patients meeting the ACR20 response criteria was assessed. A patient had an ACR20 response if all of the following occurred: A ≥ 20 % improvement in the swollen joint count (66 joints), A ≥ 20 % improvement in the tender joint count (68 joints), A ≥ 20 % improvement in at least three of the following assessments: Patient's assessment of pain, Patient's global assessment of disease activity (equivalent to the General Health component of the Disease Activity Score ([DAS]), Physician's global assessment of disease activity, Patient's assessment of physical function, as measured by the Health Assessment Questionnaire - Disability Index (HAQ-DI) Acute phase reactant (C-reactive protein [CRP]).
Time Frame: Week 48.
Population: FAS, All patients who discontinue treatment, are lost-to-follow-up or have any severe violation related to any therapy that may significantly impact efficacy assessment prior to the secondary endpoint assessment will be considered as a non-responder (NRI).
Measure: Number; unit: Percentage of patients (%)
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
Number analyzed (Participants) | 225 | 103 | 101
Percentage of patients (%) | 76.9 | 76.7 | 73.3

4. Secondary Outcome: Percentage of Patients Who Meet the American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) Definition of Remission at Week 48
Description: The ACR/EULAR remission criteria were based on a Boolean definition. At any time point, the patient must have satisfied all of the following:
  * Tender joint count (TJC) ≤ 1
  * Swollen joint count (SJC) ≤ 1
  * C-reactive protein (CRP) ≤ 1 mg/dL
  * Patient global assessment of disease activity ≤ 10 (on a 0 to 100 scale) For TJC and SJC, use of a 28-joint count may have missed actively involved joints, particularly in the feet and ankles. It was preferable to include the feet and ankles when evaluating remission.
Time Frame: Week 48.
Population: FAS
Measure: Number; unit: Percentage of patients (%)
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
Number analyzed (Participants) | 225 | 103 | 101
Percentage of patients (%) | 8.4 | 9.7 | 6.9

5. Secondary Outcome: Percentage of Patients With European League Against Rheumatism (EULAR) Response (Good Response, Moderate Response, or no Response) at Week 48
Description: Percentage of patients with European League Against Rheumatism (EULAR) response (good response, moderate response, or no response) were calculated at Week 48 for assessment of this outcome measure.
  No response: If improvement in DAS28 (ESR) at w48 <=0.6, or if DAS28(ESR) at w48 >5.1 and improvement is in range >0.6 to <1.2.
  Moderate response: If DAS28(ESR) at w48 <=5.1 and improvement is in range >0.6 to <1.2, or, DAS28(ESR) at w48 >3.2 and improvement is in range >=1.2.
  Good response: If DAS28(ESR) at w48 <=3.2 and improvement >=1.2.
Time Frame: Week 48.
Population: FAS
Measure: Number; unit: Percentage of patients (%)
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
Number analyzed (Participants) | 225 | 103 | 101
Percentage of patients (%)
  Good Response | 37.8 | 37.9 | 41.6
  Moderate Response | 49.8 | 54.4 | 51.5
  No Response | 9.3 | 5.8 | 3.0

ADVERSE EVENTS:
Time Frame: From the first drug administration until 10 weeks after the last drug administration, up to 58 weeks.
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. SAF was used for AE assessment.
Arm/Group | BI 695501 to BI 695501 | Humira® to Humira® | Humira® to BI 695501
All-Cause Mortality (participants affected / at risk) | 1/225 | 0/103 | 0/102
Serious Adverse Events (participants affected / at risk) | 14/225 | 8/103 | 4/102
Other Adverse Events (participants affected / at risk) | 9/225 | 6/103 | 2/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 to BI 695501 (N=225) | Humira® to Humira® (N=103) | Humira® to BI 695501 (N=102)
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 to BI 695501 (N=225) | Humira® to Humira® (N=103) | Humira® to BI 695501 (N=102)
Upper respiratory tract infection (Infections and infestations) | 9 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT02640612/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT02640612/SAP_001.pdf